CLINICAL TRIAL: NCT04130984
Title: Intraosseous Versus Intravenous Vascular Access During Resuscitation Following Out-of-Hospital Cardiac Arrest: A Multicenter Randomized Controlled Trial
Brief Title: Intraosseous Versus Intravenous Vascular Access During Resuscitation Following Out-of-Hospital Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); The Sixth Affiliated Hospital of Wenzhou Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Shanghai 10th People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other); Shanghai Zhongshan Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shandong Provincial Hospital (Other Government); The Third Affiliated Hospital of Wenzhou Medical University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: z2jzk20191015
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2019-10

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Out-of-Hospital Cardiac Arrest; Intraosseous; Intravenous; Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IO (Experimental): Intraosseous assess will be established in group IO, using EZ-IO for drug or fuild resuscitation. Proximal tibia is the insertion site,locating at 1 cm medial tibial tuberosity. IO access should be retained for less than 1 day, and venous access should be established as soon as possible after winning rescue time to continue treatment. Other treatment measures refer to 2015 AHA guidelines.
  Interventions: Device: EZ-IO
- Group IV (No Intervention): Intravenous access will be established in group IV, choosing any available peripheral venous for the administration of drugs or fluids.The antecubital vein is the preferred choice. If failed, the next catheterization plan will be determined by the physician in charge of the scene.Other treatment measures also refer to 2015 AHA guidelines.

INTERVENTIONS:
Device: EZ-IO — The insertion site locates at 1 cm medial tibial tuberosity. EZ-IO (U.S. Teleflex® Corporation) will be used with an adult 15G needle. Pull out the needle when having a sense of frustration, withdraw the bone marrow with the syringe, bolus 20 mL of normal saline to open intramedullary path and begin drug resuscitation at the same time. The retention time of IO route should be less than 24 h, and venous access should be established after winning rescue time as soon as possible to continue treatment.
  Other Names: IO device
  Arms: Group IO

SUMMARY:
1. Background:

   Intraosseous (IO) access is a new, fast, safe and efficient route of rescue of critically ill patients. Studies found drug pharmacokinetics and pharmacodynamics of IO are similar to IV route. Compared with IV and CVC, IO is time-consuming, easy to grasp, and has high operation success rate. Guidelines recommend IO when the establishment of vascular access is difficult or impossible.

   Recent animal studies suggest that IO access have better ventricular fibrillation termination rates, ROSC rates and survival compared with IV route. However, recent retrospective clinical studies found that IO versus IV treatment was associated with a lower likelihood of ROSC and hospitalization. How routes of vascular access influence clinical outcomes after OHCA merits multicenter randomized controlled trial. We suppose IO versus IV treatment is associated with a higher likelihood of ROSC and hospital and discharge survival.
2. Materials and methods:

   Study design This study is a prospective, open, two-arm, multicenter randomized controlled trial. The study will be conducted by 22 medical centers or affiliated hospitals in China. We will enroll nearly 2356 OHCA patients by the eligibility and exclusion criteria during January 2020 to December 2022. All of the patients will be randomized to one of 2 routes of vascular access: tibial intraosseous or peripheral intravenous. Other treatment measures of two groups refer to 2015 AHA Advanced Cardiovascular Life Support guidelines.

   Statistical analysis Intention-to-treat analysis (ITT) and per-protocol set (PPS) sensitivity analysis will be conducted in our study. Categorical variables are presented as counts and percentages, and differences are analyzed using the χ2 test. Continuous variables are presented as means with standard deviations or median (interquartile range [IQR]), and analysis is done by the Student t test or the Mann-Whitney U test according to normal or non-normal distributions.
3. Sample Size Calculation Set the following assumptions: alpha 0.025, beta 80%, clinically significant difference of 5% and 25% ROSC rate for both arms. Assuming the sample has an equal number of subjects in each arm, the study need to include at least 1178 subjects per arm to reach statistical significance.

DETAILED DESCRIPTION:
1. Background:

   Successful vascular access is critical for the treatment of acute and critically ill patients, especially those with cardiac arrest. For cardiac arrest patients, besides high-quality chest compressions and defibrillation, timely use of rescue drugs is also important. This requires early vascular access during chest compressions. Clinical studies and animal experiments indicate that 1 min delay of administration of antiarrhythmic drugs will increase the risk of adverse outcome, also found that the time interval from cardiac arrest to the first dose of rescue medication is closely related to the return of spontaneous circulation (ROSC) and prognosis.

   Because of the circulatory failure of patients with cardiac arrest, peripheral venous network often collapses, which makes it more difficult to develop vascular access. In addition, central venous catheterization (CVC) often takes an experienced physician at least 5-10 min, and it may affect resuscitation.

   Intraosseous (IO) access is a new, fast, safe and efficient route of rescue of critically ill patients. Animal and clinical studies found drug pharmacokinetics and pharmacodynamics of IO are similar to IV route. Compared with IV and CVC, IO is time-consuming, easy to grasp, and has high operation success rate. European Resuscitation Council (ERC) 2015 guidelines recommend IO when the establishment of vascular access is difficult or impossible.

   Recent animal studies suggest that IO access have better ventricular fibrillation termination rates, ROSC rates and survival compared with IV route. However, recent retrospective clinical studies found that IO versus IV treatment was associated with a lower likelihood of ROSC and hospitalization. How routes of vascular access influence clinical outcomes after OHCA merits multicenter randomized controlled trial. We suppose IO versus IV treatment is associated with a higher likelihood of ROSC and hospital and discharge survival.
2. Materials and methods:

   Study Design:

   This study is a prospective, open, two-arm, multicenter randomized controlled trial. The study will be conducted by the Department of Emergency Medicine, Second Affiliated Hospital, Zhejiang University, and other 21 medical centers or affiliated hospitals in China.

   Selection of patients:

   We will enroll nearly 2356 patients experiencing an out of hospital cardiac arrest (OHCA) patients by the eligibility and exclusion criteria during January 2020 to December 2022.

   Randomization:

   Block randomization will be conducted in this study. Randomized sequence numbers, which will be generated by the computer random number generator from Department of Medical Statistics and Epidemiology, School of Public Health, Zhejiang University, will be put into opaque envelopes and saved by an independent third party. A section included 4 random numbers, and each reference unit has its own independent research random number segment. avoiding centers into groups selectively shift caused by uneven. Research institutions and researchers should random subjects into the groups according to the random envelope numbers without secretly opening the envelope or jumping numbers. After being unpacked, random envelopes will be uniformly sealed and saved. Patients consistent with inclusion and exclusion criteria will be randomized into IO group or peripheral venous access group (IV).

   Patients will be randomized using a random envelope method, and researchers of all centers are not aware of the length of randomized block. Preparation and production of random envelops are commissioned by the Department of Emergency Medicine, Second Affiliated Hospital, Zhejiang University. The study is an open label study. But the staff responsible for the follow-up, data collection and data analysis later does not know the specific grouping. To avoid rescue delay, random envelope will be placed in fixed position in all research centers. When an OHCA patient is enrolled, randomly open a random envelope and determine the grouping.

   Intervention:

   Group IO: The insertion site locates at 1 cm medial tibial tuberosity. EZ-IO (U.S. Teleflex® Corporation) will be used with an adult 15G needle. Pull out the needle when having a sense of frustration, withdraw the bone marrow with the syringe, bolus 20 mL of normal saline to open intramedullary path and begin drug resuscitation at the same time. The retention time of IO route should be less than 24 h, and venous access should be established after winning rescue time as soon as possible to continue treatment. If failed, the next catheterization plan will be determined by the physician in charge of the scene.

   Group IV: Any available peripheral venous can be chose to establish vascular access for the administration of drugs or fluids, the antecubital vein is preferred. If failed, the next catheterization plan will be determined by the physician in charge of the scene.

   Other treatment measures of two groups refer to 2015 AHA Advanced Cardiovascular Life Support guidelines.

   Technical Training:

   The operators of IO receive at least 1 h theoretical study and practice in training until master mold puncture technique, passing the examination before the start of the study. Operators of peripheral venipuncture have more than 1 year venipuncture experience.

   Statistical analysis:

   Intention-to-treat analysis (ITT) and per-protocol set (PPS) sensitivity analysis will be conducted in our study. Descriptive statistics are used to summarize the data. Categorical variables are presented as counts and percentages, and differences between groups are analyzed using the χ2 test. Continuous variables are presented as means with standard deviations or median (interquartile range [IQR]), hence analysis is done by the Student t test or the Mann-Whitney U test according to normal or non-normal distributions. Stage analysis will be performed when collected data account for 30%, 50%, 80%, 100% of anticipation. The interim analysis will follow the O'Brien-Fleming rule to assess the safety and efficacy of this study. If the results of interim study do not meet the criteria of suspension, cases will continue to be collected until the completion of the target sample size.
3. Sample Size Calculation Prior to the start of the study a sample size calculation was performed to determine study feasibility. Model assumptions were made based on prior quality assurance reviews. Sample size requirements for a non-inferiority comparison were calculated using the following assumptions: alpha 0.025, beta 80%, clinically significant difference of 5% increase in ROSC and 25% ROSC rate for both arms. Assuming the sample has an equal number of subjects in each arm, the study would need to include at least 1178 subjects per arm (2356 total) to reach statistical significance.
4. Data Management and Confidentiality

   Data Management:

   Using EDC platform+ paper version for data management and storage. The person responsible for collecting paper version will input data in EDC platform uniformly, summary paper and electronic versions for further statistical analysis and preservation.

   Security measures:

   All records related to the identity of subjects are to be confidential and not open to the public outside the scope of relevant laws or regulations.
5. Informed consent:

   Subjects must obtain written informed consent prior to the implementation, being informed of specific content of study, as detailed informed consent.
6. Adverse events reporting:

Definition of adverse events and classification of serious adverse events:

Adverse events (AE): It is defined as any adverse medical events occurred in patients, which is not necessarily a cause or result of treatment. Therefore, adverse event can be any discomfort or unconscious signs (including abnormal laboratory findings), symptom or disease generated after interventions, whether or not considered to be related to drugs.

Serious adverse events (SAE):

Death, life-threatening, hospitalization, prolonged hospitalization, persistent or significant disability / loss of function, important medical events that require medical or surgical treatment to avoid serious consequences.

Assessment of adverse events:

In each AE, researchers need to assess: intensity (severity), clinical relevance, causality (relationship between drugs and research process), results and measures taken.

Recording and reporting procedures:

During the study, researchers should record all AE in detail and report. All SAE are required to be recorded in the AE page of CRF. In addition, a completed "serious adverse events" should be sent to the competent authorities, the local Food and Drug Administration investigators and Ethics Committee involved immediately (at the latest within 24 hours). The researcher will sign and date the report, informing the other researchers involved in this clinical study at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest patients with 18 years or more

Exclusion Criteria:

* Traumatic cardiopulmonary arrest with an indication of withholding of resuscitation, including:

  * trauma victims with injuries that are obviously incompatible with life, such as decapitation or hemicorporectomy;
  * victims of either blunt or penetrating trauma when there is evidence of prolonged cardiac arrest, including rigor mortis or dependent lividity;
  * blunt trauma patient who, on the arrival of emergency medical services (EMS) personnel, is found to be apneic, pulseless, and without organized electrocardiographic activity;
  * penetrating trauma patients who, on the arrival of EMS personnel, is found to be pulseless and apneic and there are no other signs of life, including spontaneous movement, electrocardiographic activity, and pupillary response;
* Vascular access has been established before admission;
* Return of spontaneous circulation before first attempt to establish vascular access;
* Quit resuscitation;
* Patients with contraindications of intraosseous access;

  * infection of insertion site, such as skin and soft tissue infections, osteomyelitis;
  * integrity damage of the target bone, such as fractures, artificial limbs, etc;
  * blood supply or return of the target bone is significantly affected, e.g. arteriovenous rupture;
  * burns of insertion site;
  * intraosseous attempt in same insertion site within 24 h;
  * compartment syndrome exists in same insertion site;
  * unclear anatomical structures of insertion site, such as obesity, malformations;
  * patients with severe bone diseases, such as imperfect osteogenesis, osteoporosis;
  * patients with right to left cardiac shunt (e.g. Tetralogy of Fallot, pulmonary atresia, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2356 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
return of spontaneous circulation (ROSC) | within 24 hours
  ROSC can be identified with the following three conditions: 1. arterial pulse can be reached; 2. effective ECG rhythm; 3. systolic blood pressure > 60 mmHg (1 mm Hg = 0.133 kPa);.

SECONDARY OUTCOMES:
first attempt success | within 24 hours
  refer to the initial attempted intraosseous or intravenous access is successful
overall success | within 24 hours
  including the initial attempted success and eventual attempted success after trying several times of intraosseous or intravenous access .
initial access interval | within 24 hours
  defined as the interval from arrival of first EMS vehicle on site to successful placement of an intraosseous or intravenous access.
initial epinephrine administration interval | within 24 hours
  defined as the interval from arrival of first EMS vehicle on site to administration of initial epinephrine
sustained ROSC | 24 hours
  the presence of ROSC maintain ≥ 24 h

OTHER OUTCOMES:
survival to discharge | a week
  whether OHCA patients survive to hospital discharge
survival to discharge without severe neurological impairment | a week
  defined as a CPC score of 1~2, which denotes survival with no more than moderate neurological disability with the ability to walk without assistance.
1-month survival without severe neurological impairment | 1 month
  patients who have survived for 1 month after cardiac arrest with a CPC score of 1~2
6-month survival without severe neurological impairment | 6 months
  patients who have survived for 6 months after cardiac arrest with a CPC score of 1~2
insertion-related complications | 1 day
  Whether compartment syndrome,osteomyelitis, cellulitis, skin abscesses,or some other complications occur in patients

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, Principal Investigator — Second Affiliated Hospital, Zhejiang Universitiy School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Though data that will be collected in our study are huge and multicentral, it is limited in part provinces of China, which makes it hard to apply for other centers in the world , so we do not have a plan to share IPD with other researchers.

REFERENCES:
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Petitpas F, Guenezan J, Vendeuvre T, Scepi M, Oriot D, Mimoz O. Use of intra-osseous access in adults: a systematic review. Crit Care. 2016 Apr 14;20:102. doi: 10.1186/s13054-016-1277-6. PMID 27075364
- [Background] Ong MEH, Chan YH, Oh JJ, Ngo AS. An observational, prospective study comparing tibial and humeral intraosseous access using the EZ-IO. Am J Emerg Med. 2009 Jan;27(1):8-15. doi: 10.1016/j.ajem.2008.01.025. PMID 19041528
- [Background] Kurowski A, Timler D, Evrin T, Szarpak L. Comparison of 3 different intraosseous access devices for adult during resuscitation. Randomized crossover manikin study. Am J Emerg Med. 2014 Dec;32(12):1490-3. doi: 10.1016/j.ajem.2014.09.007. Epub 2014 Sep 18. PMID 25440232
- [Background] Reades R, Studnek JR, Vandeventer S, Garrett J. Intraosseous versus intravenous vascular access during out-of-hospital cardiac arrest: a randomized controlled trial. Ann Emerg Med. 2011 Dec;58(6):509-16. doi: 10.1016/j.annemergmed.2011.07.020. PMID 21856044
- [Background] Soar J, Nolan JP, Bottiger BW, Perkins GD, Lott C, Carli P, Pellis T, Sandroni C, Skrifvars MB, Smith GB, Sunde K, Deakin CD; Adult advanced life support section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 3. Adult advanced life support. Resuscitation. 2015 Oct;95:100-47. doi: 10.1016/j.resuscitation.2015.07.016. No abstract available. PMID 26477701
- [Background] Mader TJ, Kellogg AR, Walterscheid JK, Lodding CC, Sherman LD. A randomized comparison of cardiocerebral and cardiopulmonary resuscitation using a swine model of prolonged ventricular fibrillation. Resuscitation. 2010 May;81(5):596-602. doi: 10.1016/j.resuscitation.2010.01.013. Epub 2010 Feb 21. PMID 20176434
- [Background] Zuercher M, Kern KB, Indik JH, Loedl M, Hilwig RW, Ummenhofer W, Berg RA, Ewy GA. Epinephrine improves 24-hour survival in a swine model of prolonged ventricular fibrillation demonstrating that early intraosseous is superior to delayed intravenous administration. Anesth Analg. 2011 Apr;112(4):884-90. doi: 10.1213/ANE.0b013e31820dc9ec. Epub 2011 Mar 8. PMID 21385987
- [Background] Feinstein BA, Stubbs BA, Rea T, Kudenchuk PJ. Intraosseous compared to intravenous drug resuscitation in out-of-hospital cardiac arrest. Resuscitation. 2017 Aug;117:91-96. doi: 10.1016/j.resuscitation.2017.06.014. Epub 2017 Jun 16. PMID 28629995
- [Background] Kawano T, Grunau B, Scheuermeyer FX, Gibo K, Fordyce CB, Lin S, Stenstrom R, Schlamp R, Jenneson S, Christenson J. Intraosseous Vascular Access Is Associated With Lower Survival and Neurologic Recovery Among Patients With Out-of-Hospital Cardiac Arrest. Ann Emerg Med. 2018 May;71(5):588-596. doi: 10.1016/j.annemergmed.2017.11.015. Epub 2018 Jan 6. PMID 29310869
- [Background] Clemency B, Tanaka K, May P, Innes J, Zagroba S, Blaszak J, Hostler D, Cooney D, McGee K, Lindstrom H. Intravenous vs. intraosseous access and return of spontaneous circulation during out of hospital cardiac arrest. Am J Emerg Med. 2017 Feb;35(2):222-226. doi: 10.1016/j.ajem.2016.10.052. Epub 2016 Oct 24. PMID 28288774
- [Background] Nguyen L, Suarez S, Daniels J, Sanchez C, Landry K, Redfield C. Effect of Intravenous Versus Intraosseous Access in Prehospital Cardiac Arrest. Air Med J. 2019 May-Jun;38(3):147-149. doi: 10.1016/j.amj.2019.02.005. Epub 2019 Mar 12. PMID 31122576
- [Background] Rittenberger JC, Menegazzi JJ, Callaway CW. Association of delay to first intervention with return of spontaneous circulation in a swine model of cardiac arrest. Resuscitation. 2007 Apr;73(1):154-60. doi: 10.1016/j.resuscitation.2006.07.029. Epub 2007 Jan 16. PMID 17223246
- [Background] Lapostolle F, Catineau J, Garrigue B, Monmarteau V, Houssaye T, Vecci I, Treoux V, Hospital B, Crocheton N, Adnet F. Prospective evaluation of peripheral venous access difficulty in emergency care. Intensive Care Med. 2007 Aug;33(8):1452-7. doi: 10.1007/s00134-007-0634-y. Epub 2007 Jun 7. PMID 17554524
- [Background] Lewis FR Jr. Prehospital intravenous fluid therapy: physiologic computer modelling. J Trauma. 1986 Sep;26(9):804-11. doi: 10.1097/00005373-198609000-00005. PMID 3746955
- [Background] Minville V, Pianezza A, Asehnoune K, Cabardis S, Smail N. Prehospital intravenous line placement assessment in the French emergency system: a prospective study. Eur J Anaesthesiol. 2006 Jul;23(7):594-7. doi: 10.1017/S0265021506000202. Epub 2006 Mar 1. PMID 16507183